CLINICAL TRIAL: NCT03027752
Title: The New Technique of Carotid Endarterectomy With Autoarterial Remodeling of Bifurcation of the Common Carotid Artery.
Brief Title: Pilot Study of Autoarterial Remodeling of Bifurcation of the Common Carotid Artery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: N-RICP-346
Record Dates: First submitted 2017-01-15; First posted 2017-01-23 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2016-08

CONDITIONS: Stenosis, Internal Carotid Artery
Keywords: carotid endaretectomy
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- carotid endarterectomy patch angioplasty (Active Comparator): Carotid endarterectomy with longitudinal incision carotid endarterectomy patch angioplasty
  Interventions: Procedure: Operation carotid endarterectomy with plastic of xenopericardial patch
- Carotid endarterectomy with autoarterial remodeling (Experimental): Carotid endarterectomy with autoarterial remodeling of bifurcation of the common carotid artery
  Interventions: Procedure: New method of operation сarotid endarterectomy with autoarterial remodeling of bifurcation CCA

INTERVENTIONS:
Procedure: Operation carotid endarterectomy with plastic of xenopericardial patch — Under local anesthesia Sol.Novocaini 0.25%, wires or endotracheal anesthesia using the standard access the bifurcation of the common carotid artery, internal carotid artery, isolated on identical distance external carotid artery. Common carotid artery cut then performed a longitudinal arteriotomy on the front of the anterior surface of the internal carotid artery. Under the visual control performs a sequence of endarterectomy of the internal carotid artery. Plastic arteriotomy performed patche of ksenoperikardial (Kemperiplas-Neo) treated with epoxy compounds.
  Arms: carotid endarterectomy patch angioplasty
Procedure: New method of operation сarotid endarterectomy with autoarterial remodeling of bifurcation CCA — Under local anesthesia Sol.Novocaini 0.25%, or endotracheal anesthesia using the standard access the bifurcation of the common carotid artery, internal carotid artery, isolated on identical distance external carotid artery. Carotid glomus separated and moves downward and backward bifurcation of the common carotid artery. External carotid artery is cut off at an angle of 45º from the mouth with a portion of the common carotid artery, then performed a longitudinal arteriotomy on the front of the medial surface of the internal carotid and posterior-lateral surface of the external carotid artery. Under the visual control performs a sequence of endarterectomy of the internal and external carotid arteries. The final recovery of the arteries is performed by crosslinking of their walls with each other in a side by side type between the internal and external carotid arteries 6/0 Polypropylene thread with two needles.
  Arms: Carotid endarterectomy with autoarterial remodeling

SUMMARY:
Comparison of two methods for revascularization of the bifurcation of common carotid artery: carotid endarterectomy with longitudinal incision carotid endarterectomy patch angioplasty compared with new technique of carotid endarterectomy with autoarterial remodeling of bifurcation of the common carotid artery

ELIGIBILITY:
Inclusion Criteria:

* stenotic lesions of the extracranial part of carotid arteries requiring surgical treatment according to national treatment guidelines (asymptomatic ICA stenosis more than 70% symptomatic ICA stenosis more than 65%)
* the length of the atherosclerotic plaques in the ICA than 1 cm
* personally signed Informed consent for participation in the study

Exclusion Criteria:

* Chronic heart failure III-IV functional class NYHA classification
* Chronic decompensated "lung" heart
* Decompensated diseases of endocrine organs (diabetes glycemia more than 10 mmol/l)
* Severe hepatic or renal insufficiency (bilirubin >80 mmol/l, creatinine >200 mmol/l)
* Polyvalent drug Allergy;
* Malignant tumor in the terminal stage with life expectancy of up to 6 months;
* Acute disruption of cerebral blood flow
* Extensive occlusion of the internal carotid artery.
* Exacerbation of systemic diseases.
* Pregnancy and lactation.
* The refusal of a patient to sign informed consent for participation in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Stroke or TIA | throughout 1 year
  according to the examination of neurologist

SECONDARY OUTCOMES:
Restenosis | 1 year
  The percentage narrowing of the lumen at the bifurcation of the carotid artery at 1 year after surgery according to the ultrasound
Restenosis | 6 months
  The percentage narrowing of the lumen at the bifurcation of the carotid artery at 6 months after surgery according to the ultrasound
paresis of the cranial nerve | up to 1 weeks
  Neurological status after surgical treatment according to the examination of neurologist
The linear flow velocity in the region of the carotid artery bifurcation | 3rd day
  The linear velocity of blood flow in the bifurcation of the carotid artery at 2-3 days after surgery according to the ultrasound
The linear flow velocity in the region of the carotid artery bifurcation | 6 months
  The linear velocity of blood flow in the bifurcation of the carotid artery after 6 months according to the ultrasound
The linear flow velocity in the region of the carotid artery bifurcation | 1 year
  The linear velocity of blood flow in the bifurcation of the carotid artery after 1 year according to the ultrasound
bleeding | 1 month
  30 days after surgery
Stenosis | 3rd day
  The percentage narrowing of the lumen at the bifurcation of the carotid artery at 2-3 days after surgery according to the ultrasound
Oxygenation of the brain | during the surgical intervention
  according to transcranial oximetry
Oxygenation of the brain | 6 months
  according to transcranial oximetry
Oxygenation of the brain | 1 year
  according to transcranial oximetry

CONTACTS AND LOCATIONS:
Locations (1):
- Novosibirsk Research Institute of Circulation Pathology, Novosibirsk, Russia